CLINICAL TRIAL: NCT03970564
Title: Routine Neck Ultrasound by Respiratory Physicians in the Diagnosis and Staging of Patients With Lung Cancer and Mediastinal Lymphadenopathy, a Prospective Pilot Study
Brief Title: Neck Ultrasound by Respiratory Physicians in Patients With Lung Cancer
Status: Completed | Type: Observational
Sponsor: University College Hospital Galway (Other)
Collaborators: European Respiratory Society (Other)
Responsible Party: Principal Investigator, Mohammed Ahmed, Clinical fellow, University College Hospital Galway
Other Study IDs: Version 01
Record Dates: First submitted 2019-05-29; First posted 2019-05-31 (Actual); Last update posted 2019-05-31 (Actual); Status verified 2019-05

CONDITIONS: Lung Cancer Metastatic; Nodes, Lung
Keywords: ultrasound; lymphadenopathy; lung cancer
MeSH Terms: conditions — Lymphadenopathy; Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Suspected lung cancer: Suspected and later on confirmed lung cancer with evidence of mediastinal lymphadenopathy on computerised tomography
  Interventions: Diagnostic Test: Neck ultrasound guide lymph node sampling

INTERVENTIONS:
Diagnostic Test: Neck ultrasound guide lymph node sampling — Neck ultrasound done first and lymph nodes larger than 5 mm that are technically feasible are sampled using fine needle aspiration and/or core needle biopsy

SUMMARY:
This is a study of routine neck ultrasound performed by respiratory physicians in patients with mediastinal lymphadenopathy and suspected lung cancer

DETAILED DESCRIPTION:
In the first phase of the study a respiratory physician was trained to perform neck ultrasound and needle sampling of enlarged cervical lymph nodes according to preset criteria. In the second phase patients with suspected lung cancer and enlarged mediastinal lymph nodes underwent routine neck ultrasound and enlarged cervical lymph nodes were sampled using fine needle and or core needle biopsy.

The outcomes of interest in the study were the rate of malignant cervical lymphadenopathy defined as pathological evidence of cancer in neck lymph node samples consistent with a lung primary, adequacy of needle sampling, patient reported experience assessed by a visual analogue of discomfort associated with needle neck sampling and EBUS, and the proportion of patients that had nodal upstaging

ELIGIBILITY:
Inclusion Criteria:

* Suspected and later on confirmed lung cancer
* Presence of at least one mediastinal lymph node measuring > 10 mm in short diameter on computerised Tomography

Exclusion Criteria:

* Age <18
* History any malignancy apart from non-melanomatous skin cancer
* Inability to give informed consent

Age Groups: Child, Adult, Older Adult
Study Population: Patients with suspected and later on confirmed lung cancer with evidence of enlarged mediastinal lymph node(s) measuring > 10 mm in short diameter on Computerised Tomography
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-10-21 (Actual); Primary Completion 2018-05-21 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
Adequacy of lymph node sampling | 7 days
  Presence of lymphocytes or malignant cells in biopsy samples

SECONDARY OUTCOMES:
Proportion of patients with malignant cervical lymphadenopathy | 7 days
  Presence of malignant cells consistent with lung cancer in cervical lymph node samples
Proportion of patients with nodal status upstaged | 7 days
  Defined as a change from cN2 to cN3 according to the 8th edition of the Tumour Node Metastasis TNM staging system

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Galway, Galway, Ireland

IPD SHARING:
Plan to Share IPD: No